CLINICAL TRIAL: NCT07355101
Title: Personalized Exercise Coaching to Improve Quality of Life in Pediatric IBD - FIT4IBDKids: Study Protocol
Brief Title: Personalized Exercise Coaching to Improve Quality of Life in Pediatric IBD
Acronym: FIT4IBDKids
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Max Kips, Medical student, Universiteit Antwerpen
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 7893
Record Dates: First submitted 2025-12-15; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Inflammatory Bowel Disease (IBD)
Keywords: Physical exercise; Fatigue; Children; Quality of Life; Adolescent
MeSH Terms: conditions — Inflammatory Bowel Diseases; Motor Activity; Fatigue

STUDY DESIGN:
Intervention Model Description: Children with IBD will be allocated into two groups. The first group of this study will consist of children with higher exercise habits, in particular obtaining a weekly Personal Activity Intelligence (PAI) score ≥100 at baseline. Peers in the second group will reach PAI scores <100 at baseline. The personalized metric for physical activity tracking named PAI quantifies how much physical activity per week is needed to reduce the risk of premature mortality from non-communicable diseases. PAI and objectively measured cardiorespiratory fitness (as indicated by VO2peak) are positively associated in a graded fashion. Seventy pediatric patients will be included in this trial. Children were considered eligible for inclusion aged between six and 18 years old and diagnosed with IBD (Crohn's Disease or Ulcerative Colitis) according to the European Society for Pediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN) Guidelines.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Higher exercise habits (Experimental): The first group of this study will consist of children with higher exercise habits, in particular obtaining a weekly Personal Activity Intelligence (PAI) score ≥100 at baseline. (The personalized metric for physical activity tracking named PAI quantifies how much physical activity per week is needed to reduce the risk of premature mortality from non-communicable diseases).
  Interventions: Behavioral: Intake session to define individualized physical activity goals; Behavioral: Personalized Motivational Coaching; Behavioral: 24 Week Exercise Programme
- Lower exercise habits (Active Comparator): Peers in the second group will reach PAI scores <100 at baseline. (The personalized metric for physical activity tracking named PAI quantifies how much physical activity per week is needed to reduce the risk of premature mortality from non-communicable diseases).
  Interventions: Behavioral: Intake session to define individualized physical activity goals; Behavioral: Personalized Motivational Coaching; Behavioral: 24 Week Exercise Programme

INTERVENTIONS:
Behavioral: Intake session to define individualized physical activity goals — The intake session of a 24 week exercise programme, designed by "Physical Activity on Prescription" (Bewegen Op Verwijzing), will define individualized physical activity goals in collaboration with the child, which encourages autonomy and active participation.
Behavioral: Personalized Motivational Coaching — A personalized coaching program designed by a multidisciplinary team to support physically inactive individuals in adopting a more active lifestyle. The intervention is characterized by professional guidance from a qualified and motivational coach with continuous follow-up. It is a holistic family-centered coaching trajectory for children aged six to 18 years. Its primary aim is to empower patients by equipping them with the necessary tools to actively engage in their treatment, while ensuring high-quality care as close to home as possible.
Behavioral: 24 Week Exercise Programme — A development of a 24 week tailored physical activity plan based on an initial assessment of PAI. The personalized exercise plan will be co-created with each child and their family, aiming to increase physical activity levels in a structured and supportive manner. The intervention will span a minimum duration of six months, in order to reduce the risk of drop-out and to promote long-term sustainability of behavioral change.

SUMMARY:
The primary objective of this research is to gain novel insights into the potential of physical activity in reducing fatigue, improving QoL and GI manifestations in children with IBD. The study design will be composed of two parallel groups to investigate the role of physical activity: on the one hand patients with higher exercise habits, on the other hand children with lower exercise habits. To this end, the two groups of pediatric IBD patients will undergo a 24 weeks exercise programme, adjunctive to their current treatment, quantified by a Health Smartwatch (Garmin Inc.). The primary outcomes will then be characterized by the PedsQoL-MFS, IMPACT-III, PCDAI and PUCAI questionnaires, as well as VO2-max quantification. The proposed research will confirm or refute current hypotheses about physical training suggesting an improvement in quality of life (QoL), fatigue and bowel symptoms in children with IBD. Furthermore, investigating the effectiveness on secondary outcomes including muscle strength and aerobic capacity will be a new contribution to current knowledge.

DETAILED DESCRIPTION:
A 24 week exercise programme is designed by "Physical Activity on Prescription" (Bewegen Op Verwijzing). This multidisciplinary team develops personalized coaching programs designed to support physically inactive individuals in adopting a more active lifestyle. The intervention is characterized by professional guidance from a qualified and motivational coach, the development of a tailored physical activity plan, and continuous follow-up. The team will develop a holistic family-centered coaching trajectory for children aged six to 18 years. The intake session in which individualized physical activity goals are defined in collaboration with the child, encourages autonomy and active participation. Based on this initial assessment, a personalized coaching plan will be co-created with each child and their family, aiming to increase physical activity levels in a structured and supportive manner. The intervention will span a minimum duration of six months, in order to reduce the risk of drop-out and to promote long-term sustainability of behavioral change. All participants will participate in one supervised intake session with "Physical Activity on Prescription" (Bewegen Op Verwijzing) at baseline assessment. Furthermore, the online application UZA@Home provides digital support and guidance to patients throughout their trajectory at the University Hospital of Antwerp (UZA). Its primary aim is to empower patients by equipping them with the necessary tools to actively engage in their treatment, while ensuring high-quality care as close to home as possible. Through the patient portal, individuals receive feedback on their intervention program and are able to consult appointments or access their medical records. The primary outcomes of this trial include differences in cardiorespiratory fitness (CRF), as assessed by maximal oxygen uptake (VO₂max), in addition to patient-reported outcomes measured by the IMPACT-III, PedsQoL-MFS, and the disease activity indices PCDAI and PUCAI. Secondary outcomes encompass a range of physical health parameters, including heart rate variability (HRV), muscular strength, resting blood pressure, basal metabolic rate, aerobic capacity, and body mass index (BMI). Intramural inflammation will be quantified through fecal calprotectin levels. Furthermore, disease activity will be evaluated using intestinal ultrasonography, standard endoscopic procedures (no study specific procedures, only standard of care biopsies) and the analysis of gastrointestinal mucins. All measurements will be conducted during each physical follow-up visit at the hospital, which will occur at the beginning, mid-intervention (except for endoscopy) and after the 24 week intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnose with IBD (Crohn's Disease or Ulcerative Colitis) according to the European Society for Pediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN) Guidelines.

Exclusion Criteria:

1. Diabetes Mellitus (all types, according to the American Diabetes Association (ADA))
2. Malnutrition or Failure to Thrive, suspected or confirmed
3. Children with malignancy
4. Children with an acute phase of IBD disease activity
5. Children who are too fatigued to apply
6. Children < 120 cm, as VO2 max cannot be measured
7. Physical inability to perform a cardiopulmonary exercise test (CPET)
8. Participation in organized exercise training programs in a research setting
9. Medical contra-indications for exercise

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in fatigue in children with IBD | From start to end of the adjunctive 24 weeks exercise programme to current treatment.
  This primary outcome will be characterized by a validated PedsQL™ Multidimensional Fatigue Scale (PedsQoL-MFS) questionnaire.
Change in Quality of Life in children with IBD | From start to end of the adjunctive 24 weeks exercise programme to current treatment.
  This primary outcomes will be characterized by the IMPACT-III questionnaire. IMPACT-III is a valid health-related quality of life questionnaire for pediatric patients who have an Inflammatory Bowel Disease (IBD). It was developed among children and adolescents who have IBD. The questionnaire can be administered as a self-report to individuals who have IBD. It provides a measure of patient views on aspects of their health like: physical well-being, emotional and social functioning, body Image.
Change in disease severity in children with IBD | From start to end of the adjunctive 24 weeks exercise programme to current treatment.
  This primary outcome will be characterized by the Pediatric Crohn's Disease Activity Index (PCDAI) which stratifies severity of Crohn's disease in pediatric patients or the Pediatric Ulcerative Colitis Activity Index (PUCAI) which determines severity of ulcerative colitis (UC) in pediatric patients.

SECONDARY OUTCOMES:
Heart rate variability (HRV) | From start to end of the adjunctive 24 weeks exercise programme to current treatment.
  A 24 h time-domain measures of SDNN (standard deviation of the IBI of normal sinus beats).
Muscular strength | From start to end of the adjunctive 24 weeks exercise programme to current treatment.
  Objective grading by Handheld Dynamometers (HHDs) to provide a precise and numerical measure of muscle force, displaying the result in quantifiable units like Newtons or kilograms.
Resting blood pressure | From start to end of the adjunctive 24 weeks exercise programme to current treatment.
  In resting conditions, systolic over diastolic blood pressure in mmHg.
Body mass index (BMI) | From start to end of the adjunctive 24 weeks exercise programme to current treatment.
  Expressed in units of kg/m2, resulting from mass in kilograms (kg) and height in metres (m).
Maximal oxygen uptake (VO₂max) | From start to end of the adjunctive 24 weeks exercise programme to current treatment.
  V̇O2max is expressed as a relative rate in (for example) millilitres of oxygen per kilogram of the body mass per minute (e.g., mL/(kg·min)).
Intestinal ultrasonograph | From start to end of the adjunctive 24 weeks exercise programme to current treatment.
  The ultrasonographic evaluation of the small and large bowels should be performed with both low-frequency (2-5 MHz) and high-frequency (5-17 MHz) linear array probes to provide a correct assessment of the bowel wall thickness and discrimination of the five different bowel wall layers (lumen/mucosa interface, mucosa, submucosa, muscolaris propria, serosa).
Standard endoscopic procedure | From start to end of the adjunctive 24 weeks exercise programme to current treatment.
  According Position Paper on Behalf of the IBD Group of the European Society for Pediatric Gastroenterology,
  Hepatology and Nutrition:
  1. Pediatric Endoscopy should be performed by a pediatric gastroenterologist, or in some cases, by a gastroenterologist with specific pediatric training and/or supported by a pediatric team in a pediatric-friendly setting, as described in the recent ESPGHAN/European Society for Gastrointestinal Endoscopy (ESGE) guidelines.
  2. According to the revised Porto Criteria, endoscopy is usually recommended in the presence of alarming symptoms (ie, bloody diarrhea, weight loss, abdominal pain) and/or positive serum inflammatory markers (C-CRP) an/or ESR), and/or high levels of fecal calprotectin.
  3. It is recommended to collect 2 biopsies samples from duodenum, stomach and esophagus during EGD, and from terminal ileum, cecum, transverse colon, sigmoid colon, and rectum during IC.
  4. In severe acute colitis, a limited sigmoidoscopy may be safer.
Fecal calprotectin level | From start to end of the adjunctive 24 weeks exercise programme to current treatment.
  Expressed in μg/g of faeces.
Gastrointestinal mucins | From start to end of the adjunctive 24 weeks exercise programme to current treatment.
  GWAS for mucin genes including MUC3A, MUC3B, MUC12, and MUC17.

CONTACTS AND LOCATIONS:
Overall Officials: Els Van de Vijver, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Edegem, Antwerpen, Belgium

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared. All anonymous data will be collected prospectively in REDCap (Research Electronic Data Capture) during scheduled hospital visits at baseline, throughout the intervention period (one follow-up point), and at study completion. Patient-reported outcomes will be obtained through validated questionnaires (IMPACT-III, PedsQoL-MFS, PCDAI, and PUCAI), administered electronically in the UZA@Home application. All data will be entered into a secure, password-protected electronic database compliant with GDPR and institutional data protection policies. Any discrepancies or missing values will be addressed according to a predefined data management plan. The four researchers adhere to the 'Guide on Good Data Protection Practice in Research' of the European University Institute (EUI). Technical appendix, statistical code, and dataset available from the Dryad repository.

REFERENCES:
- [Background] Cozijnsen MA, van Pieterson M, Samsom JN, Escher JC, de Ridder L. Top-down Infliximab Study in Kids with Crohn's disease (TISKids): an international multicentre randomised controlled trial. BMJ Open Gastroenterol. 2016 Dec 22;3(1):e000123. doi: 10.1136/bmjgast-2016-000123. eCollection 2016. PMID 28090335
- [Background] Bishop J, Lemberg DA, Day A. Managing inflammatory bowel disease in adolescent patients. Adolesc Health Med Ther. 2014 Jan 6;5:1-13. doi: 10.2147/AHMT.S37956. eCollection 2014. PMID 24729736
- [Background] Arruda JM, Bogetz AL, Vellanki S, Wren A, Yeh AM. Yoga as adjunct therapy for adolescents with inflammatory bowel disease: A pilot clinical trial. Complement Ther Med. 2018 Dec;41:99-104. doi: 10.1016/j.ctim.2018.09.007. Epub 2018 Sep 11. PMID 30477870
- [Background] Legeret C, Mahlmann L, Gerber M, Kalak N, Kohler H, Holsboer-Trachsler E, Brand S, Furlano R. Favorable impact of long-term exercise on disease symptoms in pediatric patients with inflammatory bowel disease. BMC Pediatr. 2019 Aug 27;19(1):297. doi: 10.1186/s12887-019-1680-7. PMID 31455308
- [Background] Scheffers LE, Vos IK, Utens EMWJ, Dieleman GC, Walet S, Escher JC, van den Berg LEM; Rotterdam Exercise Team. Physical Training and Healthy Diet Improved Bowel Symptoms, Quality of Life, and Fatigue in Children With Inflammatory Bowel Disease. J Pediatr Gastroenterol Nutr. 2023 Aug 1;77(2):214-221. doi: 10.1097/MPG.0000000000003816. Epub 2023 May 3. PMID 37134004
- [Background] Mackner LM, Greenley RN, Szigethy E, Herzer M, Deer K, Hommel KA. Psychosocial issues in pediatric inflammatory bowel disease: report of the North American Society for Pediatric Gastroenterology, Hepatology, and Nutrition. J Pediatr Gastroenterol Nutr. 2013 Apr;56(4):449-58. doi: 10.1097/MPG.0b013e3182841263. PMID 23287808
- [Background] Greenley RN, Hommel KA, Nebel J, Raboin T, Li SH, Simpson P, Mackner L. A meta-analytic review of the psychosocial adjustment of youth with inflammatory bowel disease. J Pediatr Psychol. 2010 Sep;35(8):857-69. doi: 10.1093/jpepsy/jsp120. Epub 2010 Feb 1. PMID 20123705
- [Background] Shaw SY, Blanchard JF, Bernstein CN. Association between the use of antibiotics in the first year of life and pediatric inflammatory bowel disease. Am J Gastroenterol. 2010 Dec;105(12):2687-92. doi: 10.1038/ajg.2010.398. Epub 2010 Oct 12. PMID 20940708
- [Background] Hou JK, Abraham B, El-Serag H. Dietary intake and risk of developing inflammatory bowel disease: a systematic review of the literature. Am J Gastroenterol. 2011 Apr;106(4):563-73. doi: 10.1038/ajg.2011.44. PMID 21468064
- [Background] Bager P, Simonsen J, Nielsen NM, Frisch M. Cesarean section and offspring's risk of inflammatory bowel disease: a national cohort study. Inflamm Bowel Dis. 2012 May;18(5):857-62. doi: 10.1002/ibd.21805. Epub 2011 Jul 7. PMID 21739532
- [Background] Kugathasan S, Judd RH, Hoffmann RG, Heikenen J, Telega G, Khan F, Weisdorf-Schindele S, San Pablo W Jr, Perrault J, Park R, Yaffe M, Brown C, Rivera-Bennett MT, Halabi I, Martinez A, Blank E, Werlin SL, Rudolph CD, Binion DG; Wisconsin Pediatric Inflammatory Bowel Disease Alliance. Epidemiologic and clinical characteristics of children with newly diagnosed inflammatory bowel disease in Wisconsin: a statewide population-based study. J Pediatr. 2003 Oct;143(4):525-31. doi: 10.1067/s0022-3476(03)00444-x. PMID 14571234
- [Background] Muise AM, Snapper SB, Kugathasan S. The age of gene discovery in very early onset inflammatory bowel disease. Gastroenterology. 2012 Aug;143(2):285-8. doi: 10.1053/j.gastro.2012.06.025. Epub 2012 Jun 21. No abstract available. PMID 22727850
- [Background] Knights D, Lassen KG, Xavier RJ. Advances in inflammatory bowel disease pathogenesis: linking host genetics and the microbiome. Gut. 2013 Oct;62(10):1505-10. doi: 10.1136/gutjnl-2012-303954. PMID 24037875
- [Background] Khor B, Gardet A, Xavier RJ. Genetics and pathogenesis of inflammatory bowel disease. Nature. 2011 Jun 15;474(7351):307-17. doi: 10.1038/nature10209. PMID 21677747
- [Background] van Rheenen PF, Aloi M, Assa A, Bronsky J, Escher JC, Fagerberg UL, Gasparetto M, Gerasimidis K, Griffiths A, Henderson P, Koletzko S, Kolho KL, Levine A, van Limbergen J, Martin de Carpi FJ, Navas-Lopez VM, Oliva S, de Ridder L, Russell RK, Shouval D, Spinelli A, Turner D, Wilson D, Wine E, Ruemmele FM. The Medical Management of Paediatric Crohn's Disease: an ECCO-ESPGHAN Guideline Update. J Crohns Colitis. 2021 Feb 1;15(2):jjaa161. doi: 10.1093/ecco-jcc/jjaa161. Epub 2020 Oct 7. PMID 33026087
- [Background] Benchimol EI, Fortinsky KJ, Gozdyra P, Van den Heuvel M, Van Limbergen J, Griffiths AM. Epidemiology of pediatric inflammatory bowel disease: a systematic review of international trends. Inflamm Bowel Dis. 2011 Jan;17(1):423-39. doi: 10.1002/ibd.21349. PMID 20564651
- [Background] Adamiak T, Walkiewicz-Jedrzejczak D, Fish D, Brown C, Tung J, Khan K, Faubion W Jr, Park R, Heikenen J, Yaffee M, Rivera-Bennett MT, Wiedkamp M, Stephens M, Noel R, Nugent M, Nebel J, Simpson P, Kappelman MD, Kugathasan S. Incidence, clinical characteristics, and natural history of pediatric IBD in Wisconsin: a population-based epidemiological study. Inflamm Bowel Dis. 2013 May;19(6):1218-23. doi: 10.1097/MIB.0b013e318280b13e. PMID 23528339
- [Background] Conrad MA, Rosh JR. Pediatric Inflammatory Bowel Disease. Pediatr Clin North Am. 2017 Jun;64(3):577-591. doi: 10.1016/j.pcl.2017.01.005. PMID 28502439
- [Background] Rosen MJ, Dhawan A, Saeed SA. Inflammatory Bowel Disease in Children and Adolescents. JAMA Pediatr. 2015 Nov;169(11):1053-60. doi: 10.1001/jamapediatrics.2015.1982. PMID 26414706

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2026-01-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT07355101/Prot_SAP_000.pdf